CLINICAL TRIAL: NCT06606236
Title: Neuropeptide Y Regulates Tooth Bleaching Agent-induced Neurogenic Pulp Inflammation: An In-Vivo Study
Brief Title: Neuropeptide Y Regulates Neurogenic Pulp Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institucion Universitaria Colegios de Colombia (Other)
Responsible Party: Principal Investigator, Javier Caviedes-Bucheli, Principal Investigator, Institucion Universitaria Colegios de Colombia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BIO407
Record Dates: First submitted 2024-09-14; First posted 2024-09-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Neurogenic Inflammation; Dental Pulp Disease
Keywords: NPY; Dental Pulp; Dental Bleaching; Neurogenic Inflammation
MeSH Terms: conditions — Neurogenic Inflammation; Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: Sample Collection:
  Teeth were anesthetized after tooth bleaching using 3% mepivacaine without a vasoconstrictor for maxillary premolars and an inferior alveolar nerve block for mandibular premolars. 10 minutes later, teeth were extracted within 5 minutes. For the control group, extractions also occurred ten minutes post-anesthesia. After extraction, teeth were rinsed with 5.25% sodium hypochlorite to eliminate any remaining periodontal ligament. Teeth were sectioned with a Zekrya bur, and pulp tissue was collected with a sterile excavator, placed in a 1 ml 4% paraformaldehyde Eppendorf tube, and stored at -70°C.
  ELISA:
  Fifty microliters of each standard, blank, and sample were added to wells in duplicate. A working solution with biotinylated antibody was added, and the plate was incubated at 37°C. After washing, horseradish peroxidase-conjugated solution was added, followed by substrate and stop solution. The optical density of each well was measured at 450 nm.
Who Masked: Investigator
Masking Description: The bleaching agent was applied using specific devices, with only the laboratory staff able to identify the corresponding group codes, which consisted of letters and numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): The teeth were not exposed to dental bleaching agents (healthy pulps with normal/basal NPY values). n=10
- Pola Office system group (Experimental): Application of Pola office n=10
  Interventions: Other: H2O2 at 35% for 8 minutes
- Opalescent Boost system group (Experimental): Application of Opalescent Boost n=10
  Interventions: Other: H2O2 at 40% for 20 minutes
- Zoom system group (Experimental): Application of Zoom! n=10
  Interventions: Other: H2O2 at 25% plus cold blue light for 15 minutes

INTERVENTIONS:
Other: H2O2 at 35% for 8 minutes — The investigators rigorously followed the manufacturer's instructions for all bleaching systems.
  Arms: Pola Office system group
Other: H2O2 at 40% for 20 minutes — The investigators rigorously followed the manufacturer's instructions for all bleaching systems.
  Arms: Opalescent Boost system group
Other: H2O2 at 25% plus cold blue light for 15 minutes — The investigators rigorously followed the manufacturer's instructions for all bleaching systems.
  Arms: Zoom system group

SUMMARY:
Objective. This study assessed the neuropeptide Y (NPY) expression in healthy human dental pulp following tooth bleaching with three in-office hydrogen peroxide-based systems: Opalescence Boost© (Ultradent Products, South Jordan, UT), Pola Office© (SDI, Victoria, Australia), and Zoom© (Zoom! Bleaching System; Discuss Dental, Culver City, CA).

Materials and Methods. Forty dental pulps were collected from healthy premolars scheduled for extraction for orthodontic reasons. Teeth were divided into four groups containing ten healthy premolars each: Control group (n= 10): the teeth were not exposed to dental bleaching agents (healthy pulps assessed for normal/basal NPY values). Pola Office system group (n= 10): application of Pola office (35% H2O2) for 8 minutes. Opalescent Boost system group (n= 10): application of Opalescent Boost (40% H2O2) for 20 minutes. Zoom system group (n= 10): application of Zoom! (25% H2O2 + cold blue light) for 15 minutes. The investigators rigorously followed the manufacturer's instructions for all bleaching systems. Following the extractions, the pulpal tissue was collected, placed in a 4% formaldehyde solution in Eppendorf tubes, and processed. NPY levels were measured using enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Dental pulps were collected from non-smoking donors
* Patients who need premolar extractions for orthodontic purposes.
* These premolars must meet the following requirements:
* Caries and restoration-free,
* Complete root development (visually and radiographically confirmed),
* Normal response to sensitivity testing.

Exclusion Criteria:

* Evidence of periodontal disease,
* Traumatic occlusion
* Previous orthodontic force application.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Neuropeptide Y expression | 8-20 minutes
  Measurement of the increase or not of NPY expression compared to the control group (teeth without intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Odontologia, Unicoc, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basting RT, Amaral FL, Franca FM, Florio FM. Clinical comparative study of the effectiveness of and tooth sensitivity to 10% and 20% carbamide peroxide home-use and 35% and 38% hydrogen peroxide in-office bleaching materials containing desensitizing agents. Oper Dent. 2012 Sep-Oct;37(5):464-73. doi: 10.2341/11-337-C. Epub 2012 May 18. PMID 22616927
- [Background] Bharti R, Wadhwani K. Spectrophotometric evaluation of peroxide penetration into the pulp chamber from whitening strips and gel: An in vitro study. J Conserv Dent. 2013 Mar;16(2):131-4. doi: 10.4103/0972-0707.108192. PMID 23716964
- [Background] Buchalla W, Attin T. External bleaching therapy with activation by heat, light or laser--a systematic review. Dent Mater. 2007 May;23(5):586-96. doi: 10.1016/j.dental.2006.03.018. Epub 2006 Jul 3. PMID 16820199
- [Background] Caviedes-Bucheli J, Munoz HR, Azuero-Holguin MM, Ulate E. Neuropeptides in dental pulp: the silent protagonists. J Endod. 2008 Jul;34(7):773-88. doi: 10.1016/j.joen.2008.03.010. PMID 18570980
- [Background] Caviedes-Bucheli J, Ariza-Garcia G, Restrepo-Mendez S, Rios-Osorio N, Lombana N, Munoz HR. The effect of tooth bleaching on substance P expression in human dental pulp. J Endod. 2008 Dec;34(12):1462-5. doi: 10.1016/j.joen.2008.09.013. Epub 2008 Oct 31. PMID 19026874
- [Background] Caviedes-Bucheli J, Gomez-Sosa JF, Azuero-Holguin MM, Ormeno-Gomez M, Pinto-Pascual V, Munoz HR. Angiogenic mechanisms of human dental pulp and their relationship with substance P expression in response to occlusal trauma. Int Endod J. 2017 Apr;50(4):339-351. doi: 10.1111/iej.12627. Epub 2016 Apr 2. PMID 26953220
- [Background] Caviedes-Bucheli J, Lombana N, Azuero-Holguin MM, Munoz HR. Quantification of neuropeptides (calcitonin gene-related peptide, substance P, neurokinin A, neuropeptide Y and vasoactive intestinal polypeptide) expressed in healthy and inflamed human dental pulp. Int Endod J. 2006 May;39(5):394-400. doi: 10.1111/j.1365-2591.2006.01093.x. PMID 16640639
- [Background] Caviedes-Bucheli J, Lopez-Moncayo LF, Munoz-Alvear HD, Hernandez-Acosta F, Pantoja-Mora M, Rodriguez-Guerrero AS, Lopez-Ordonez A, Diaz LE, Gomez-Sosa JF, Munoz HR. Expression of early angiogenesis indicators in mature versus immature teeth. BMC Oral Health. 2020 Nov 12;20(1):324. doi: 10.1186/s12903-020-01313-1. PMID 33183306
- [Background] Donato MV, Dos Reis-Prado AH, Abreu LG, de Arantes LC, Goto J, Chaves HGDS, Cintra LTA, Briso ALF, Peixoto IFDC, Benetti F. Influence of dental bleaching on the pulp tissue: A systematic review of in vivo studies. Int Endod J. 2024 Jun;57(6):630-654. doi: 10.1111/iej.14061. Epub 2024 Mar 12. PMID 38470103
- [Background] El-Karim I, Lundy FT, Linden GJ, Lamey PJ. Extraction and radioimmunoassay quantitation of neuropeptide Y (NPY) and vasoactive intestinal polypeptide (VIP) from human dental pulp tissue. Arch Oral Biol. 2003 Mar;48(3):249-54. doi: 10.1016/s0003-9969(02)00213-3. PMID 12648563
- [Background] Farah RI, Elwi H. Spectrophotometric evaluation of color changes of bleach-shade resin-based composites after staining and bleaching. J Contemp Dent Pract. 2014 Sep 1;15(5):587-94. doi: 10.5005/jp-journals-10024-1584. PMID 25707831
- [Background] Fernandes AMM, Vilela PGF, Valera MC, Bolay C, Hiller KA, Schweikl H, Schmalz G. Effect of bleaching agent extracts on murine macrophages. Clin Oral Investig. 2018 May;22(4):1771-1781. doi: 10.1007/s00784-017-2273-1. Epub 2017 Dec 1. PMID 29196947
- [Background] Galler KM, Weber M, Korkmaz Y, Widbiller M, Feuerer M. Inflammatory Response Mechanisms of the Dentine-Pulp Complex and the Periapical Tissues. Int J Mol Sci. 2021 Feb 2;22(3):1480. doi: 10.3390/ijms22031480. PMID 33540711